CLINICAL TRIAL: NCT01663480
Title: Assessment of Patient-ventilator Breath Contribution (PVBC) During Neurally Adjusted Ventilatory Assist (NAVA) in Patients With Acute Respiratory Failure
Brief Title: To Identify the Proportionality of Respiratory Work Under Different NAVA Level
Status: Completed | Type: Observational
Sponsor: Ling Liu (Other)
Responsible Party: Sponsor-Investigator, Ling Liu, professor, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: NAVA3
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of mechanical ventilation is to sufficiently unload the respiratory muscles and maintain adequate ventilation in spontaneously breathing patients. When the mechanical ventilatory assist is synchronized to the patient's inspiratory effort, both the patient and the mechanical ventilator will contribute to the lung-distending pressure, necessary to overcome inspiratory load and generate the tidal volume (Vt). Unfortunately, conventional modes of mechanical ventilation cannot quantify the impact of the ventilatory assist performed by the ventilator and the patient. Inadequate levels of assist are associated with adverse effects such as development of fatigue or patient-ventilator dissynchrony and diaphragm impairment, and over assist also lead to diaphragm atrophy and weaning delay.

The newly introduced neurally adjusted ventilatory assist (NAVA) has made it possible to measure the neural activity of the respiratory centers (expressed by the diaphragm electrical activity, EAdi). EAdi is a validated variable to quantify the neural respiratory drive, little is known about its usefulness to evaluate the contribution of the patient's inspiratory muscle effort relative to that of the mechanical ventilator, which would be of crucial importance to appropriately titrate the level of assist.

During NAVA, the patient's efficiency to transform neural effort (EAdi) into Vt, expressed as neuroventilatory efficiency (NVE), may be a useful predictor for determining the contribution of the patient and the ventilator to generate a breath.

ELIGIBILITY:
Inclusion Criteria:(1) Intubated or tracheostomied patients with ARF due to COPD (10 patients) or other reasons (10 patients) who were undergoing assisted mechanical ventilation, (2) be able to tolerate short time (30 minutes) spontaneous breathing (PEEP≤5cmH2O, without assist), (3) awake and do not need high dose of sedation

Exclusion Criteria:(1) age <18 or >80 years, (2) ready for extubation, (3) history of esophageal varices, (4) gastro-esophageal surgery in the previous 12 months or gastro-esophageal bleeding in the previous 30 days, (5) coagulation disorders (INR ratio>1.5 and APTT>44 s), (6) history of acute central or peripheral nervous system disorder or severe neuromuscular disease, (7) history of leukemia, severe chronic liver or chronic cardiac disease, (8) solid organ transplantation, (9) malignant tumor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with respiratery failure need mechinical ventilation, and will be tolerance short time loe level support ventilation
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
PVBC index | every 3 mins
  PVBC2predicts the contribution of the inspiratory muscles versus that of the ventilator during NAVA

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, Study Director — southeast univerity, China
Locations (1):
- Southeast Univerity, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Liu L, Liu S, Xie J, Yang Y, Slutsky AS, Beck J, Sinderby C, Qiu H. Assessment of patient-ventilator breath contribution during neurally adjusted ventilatory assist in patients with acute respiratory failure. Crit Care. 2015 Feb 18;19(1):43. doi: 10.1186/s13054-015-0775-2. PMID 25882607